CLINICAL TRIAL: NCT00525824
Title: A 12-week Open-label, Randomised, Parallel-group, Multicentre, Phase IIIb Study to Compare the Efficacy and Safety of Rosuvastatin (CRESTOR™) in Combination With Ezetimibe and Simvastatin in Patients With Hypercholesterolaemia and CHD
Brief Title: 12-week Open-label, Phase IIIb Comparing Efficacy and Safety of Rosuvastatin (CRESTOR™) in Combination With Ezetimibe
Acronym: GRAVITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Michael Cressman - Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D356FC00003
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Results first posted 2009-10-07 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease; Atherosclerosis
Keywords: Hypercholesterolaemia; Coronary Heart Disease (CHD); Atherosclerosis
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease; Atherosclerosis | interventions — Rosuvastatin Calcium; Ezetimibe; Simvastatin

INTERVENTIONS:
Drug: Rosuvastatin (Crestor) — 10mg and 20 mg
Drug: Ezetimibe — 10 mg
Drug: Simvastatin — 40mg and 80 mg

SUMMARY:
The purpose of this study is to determine whether treatment of Rosuvastatin (CRESTOR™) or Simvastatin given as monotherapy or given in combination with Ezetimibe, will lower the Low Density Lipoprotein Cholesterol (LDL-C) in patients with Hypercholesterolaemia and Coronary Heart Disease (CHD) or a CHD Risk Equivalent, Atherosclerosis or a 10-year CHD Risk of >20%

ELIGIBILITY:
Inclusion Criteria:

* Patients with with hypercholesterolaemia and CHD or a CHD risk equivalent, clinical evidence of atherosclerosis or a Framingham 10-year CHD risk score of >20
* Patients will need to sign an informed consent before any visit procedures can be performed, including procedures for the optional genetic research and biomarker studies.
* Patients must be 18 years or older and will be asked to stop taking any current cholesterol-lowering medications. Dietary counselling will be provided which will include an overview of the Therapeutic Lifestyle Change (TLC) diet the patients will be asked to follow

Exclusion Criteria:

* Use of lipid lowering drugs and other prohibited concomitant medications. History of statin-induced myopathy, or serious hypersensitivity reaction to other HMG-CoA reductase inhibitors (statins), including rosuvastatin, simvastatin and/or a history of hypersensitivity to any components of ezetimibe.
* Patients considered to be unstable by their physician after the following events:

a myocardial infarction, recent episode of unstable angina, myocardial revascularisation [percutaneous transluminal coronary angioplasty (PTCA), coronary artery bypass graft (CABG) surgery or another revascularisation procedure] or a transient ischaemic attack (TIA) or stroke and patients awaiting a planned myocardial revascularisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1743 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christie M Ballantyne, MD FACP FACC, Principal Investigator — Centre for Cardiovascular Disease Prevention; Margareta Grind, MD PhD FFPM, Study Chair — Medicine and Sciences AstraZeneca
Locations (9):
- Research Site, Brentwood, Tennessee, United States
- Research Site, Buenos Aires, Argentina
- Research Site, São Paulo, São Paulo, Brazil
- Research Site, Santiago, Chile
- Research Site, Brentwood, Colombia
- Research Site, Brentwood, Lithuania
- Research Site, Zwinderen, Netherlands
- Research Site, Lima, San Isidro Lima, Peru
- Research Site, Brentwood, Venezuela

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight hundred thirty-three patients (with hypercholesterolaemia and CHD or CHD risk equivalent, atherosclerosis or a 10-year CHD risk of >20%) were randomized into the study, from 111 sites located in the United States (56), Peru (13), Netherlands (12), Colombia (8), Argentina (8), Brazil (6), Chile (4) and Lithuania (4).
Pre-assignment Details: Patients underwent screening procedures (Week -6; Visit 1), and entered a 6-week dietary lead-in period. Those who fulfilled all eligibility criteria (Week -6; Visit 1) and had qualifying lipid values at Visit 2 were randomly allocated (1:1:1:1) to 1 of 4 treatments for a period of 12 weeks.
Groups:
- R10 to R10 + E10: Rosuvastatin 10 mg followed by Rosuvastatin 10 mg + Ezetimibe 10 mg
- R20 to R20 + E10: Rosuvastatin 20 mg followed by Rosuvastatin 20 mg + Ezetimibe 10 mg
- S40 to S40 + E10: Simvastatin 40 mg followed by Simvastatin 40 mg + Ezetimibe 10 mg
- S80 to S80 + E10: Simvastatin 80 mg followed by Simvastatin 80 mg + Ezetimibe 10 mg
Period: Overall Study
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Started | 214 (Randomized population) | 214 (Randomized population) | 202 (Randomized population) | 203 (Randomized population)
Completed | 195 | 186 | 183 | 188
Not Completed | 19 | 28 | 19 | 15
Not completed — Adverse Event | 7 | 11 | 6 | 7
Not completed — Withdrawal by Subject | 5 | 9 | 3 | 4
Not completed — Lost to Follow-up | 4 | 2 | 4 | 0
Not completed — Incorrect enrolment/mis-randomisation | 1 | 2 | 1 | 2
Not completed — Severe non-compliance | 0 | 1 | 1 | 1
Not completed — Safety reasons | 1 | 0 | 1 | 0
Not completed — Other | 1 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10 | Total
Number analyzed (Participants) | 214 | 214 | 202 | 203 | 833
Age Continuous [Mean (Standard Deviation); unit: years] | 62.2 (10.14) | 61.8 (9.93) | 61.9 (9.37) | 62.1 (9.17) | 62.0 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91.0000 | 97.0000 | 97.0000 | 90.0000 | 375.0
  Male | 123.0000 | 117.0000 | 105.0000 | 113.0000 | 458.0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) After 6 Weeks Combination Treatment
Description: Percent change in LDL-C = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 210 | 204 | 199 | 201
Percentage | -59.7200 (14.1660) | -63.4800 (16.6970) | -55.2200 (15.7500) | -57.4200 (20.4660)

2. Secondary Outcome: Percent Change in High-density Lipoprotein Cholesterol (HDL-C) After 6 Weeks Combination Treatment
Description: Percent change in HDL-C = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 210 | 204 | 199 | 201
Percentage | 6.4100 (13.9340) | 7.4600 (16.3510) | 3.9200 (12.6830) | 4.3400 (12.6430)

3. Secondary Outcome: Percent Change in Total Cholesterol (TC) After 6 Weeks Combination Treatment
Description: Percent change in TC = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 210 | 204 | 199 | 201
Percentage | -43.0000 (11.2080) | -46.6300 (12.8180) | -39.5600 (12.6640) | -41.7100 (15.1500)

4. Secondary Outcome: Percent Change in Triglycerides (TG) After 6 Weeks Combination Treatment
Description: Percent change in TG = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 210 | 204 | 199 | 201
Percentage | -28.8500 (23.7090) | -35.0000 (23.9710) | -22.9500 (28.1390) | -25.8200 (26.6190)

5. Secondary Outcome: Percent Change in Non-high-density Lipoprotein Cholesterol (nonHDL-C) After 6 Weeks Combination Treatment
Description: Percent change in nonHDL-C = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 210 | 204 | 199 | 201
Percentage | -54.6500 (13.6770) | -58.9100 (14.9320) | -49.9300 (14.7380) | -52.3700 (18.4290)

6. Secondary Outcome: Percent Change in Apolipoprotein B (ApoB) After 6 Weeks Combination Treatment
Description: Percent change in ApoB = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 206 | 199 | 194 | 199
Percentage | -46.1100 (12.6280) | -49.5000 (13.8210) | -41.9500 (14.7500) | -44.1700 (17.1790)

7. Secondary Outcome: Percent Change in Apolipoprotein A1 (ApoA-1) After 6 Weeks Combination Treatment
Description: Percent change in ApoA-1 = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 206 | 199 | 194 | 199
Percentage | 3.8100 (13.0420) | 2.6800 (11.5020) | 1.4900 (9.6830) | 2.1300 (10.7410)

8. Secondary Outcome: Percent Change in TC/HDL-C After 6 Weeks Combination Treatment
Description: Percent change in TC/HDL-C = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 210 | 204 | 199 | 201
Percentage | -45.5200 (13.2280) | -49.4600 (13.5750) | -41.2700 (13.0210) | -43.4500 (16.3430)

9. Secondary Outcome: Percent Change in LDL-C/HDL-C After 6 Weeks Combination Treatment
Description: Percent change in LDL-C/HDL-C = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 210 | 204 | 199 | 201
Percentage | -61.4700 (15.5470) | -65.2500 (16.6800) | -57.1300 (14.7770) | -58.6600 (21.1300)

10. Secondary Outcome: Percent Change in Non-HDL-C/HDL-C After 6 Weeks Combination Treatment
Description: Percent change in non-HDL-C/HDL-C = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 210 | 204 | 199 | 201
Percentage | -56.4200 (15.4150) | -60.8900 (15.5030) | -51.1100 (15.3800) | -53.5100 (20.2230)

11. Secondary Outcome: Percent Change in ApoB/ApoA-1 After 6 Weeks Combination Treatment
Description: Percent change in ApoB/ApoA-1 = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 206 | 199 | 194 | 199
Percentage | -47.3900 (13.8690) | -50.2400 (14.2570) | -42.5400 (14.2480) | -44.7600 (17.8420)

12. Secondary Outcome: Percent Change in High-sensitivity C-reactive Protein (Hs-CRP) After 6 Weeks Combination Treatment
Description: Percent change in hs-CRP = (Combination treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on combination therapy (Last observation carried forward)
Measure: Mean (Full Range); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 207 | 202 | 197 | 199
Percentage | 107.1200 (-99.0000) [-99.0 to 20295.0] | -9.5300 (-97.9000) [-97.9 to 2368.3] | 15.0300 (-91.5000) [-91.5 to 1611.4] | 0.4200 (-94.9000) [-94.9 to 1270.4]

13. Secondary Outcome: Percent Change in LDL-C After 6 Weeks Monotherapy
Description: Percent change in LDL-C = (Monotherapy treatment value - Baseline value)/Baseline value*100
Time Frame: Mean of Weeks 4 and 6 on monotherapy (Last observation carried forward)
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | R10 to R10 + E10 | R20 to R20 + E10 | S40 to S40 + E10 | S80 to S80 + E10
Number analyzed (Participants) | 206 | 199 | 197 | 200
Percentage | -46.4900 (13.1080) | -53.5900 (10.5030) | -40.8600 (12.4130) | -46.3500 (16.1880)

ADVERSE EVENTS:
Groups:
- Rosuvastatin 10 mg: Rosuvastatin 10 mg Monotherapy arm
- Rosuvastatin 20 mg: Rosuvastatin 20 mg Monotherapy arm
- Simvastatin 40 mg: Simvastatin 40 mg Monotherapy arm
- Simvastatin 80 mg: Simvastatin 80 mg Monotherapy arm
- Rosu 10 mg + Eze 10 mg: Rosuvastatin 10 mg + Ezetimibe 10 mg
- Rosu 20 mg + Eze 10 mg: Rosuvastatin 20 mg + Ezetimibe 10 mg
- Simva 40 mg + Eze 10 mg: Simvastatin 40 mg + Ezetimibe 10 mg
- Simva 80 mg + Eze 10 mg: Simvastatin 80 mg + Ezetimibe 10 mg
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Simvastatin 40 mg | Simvastatin 80 mg | Rosu 10 mg + Eze 10 mg | Rosu 20 mg + Eze 10 mg | Simva 40 mg + Eze 10 mg | Simva 80 mg + Eze 10 mg
Serious Adverse Events (participants affected / at risk) | 3 | 5 | 1 | 3 | 4 | 1 | 7 | 4
Other Adverse Events (participants affected / at risk) | 25 | 31 | 28 | 26 | 18 | 23 | 24 | 21
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Simvastatin 40 mg | Simvastatin 80 mg | Rosu 10 mg + Eze 10 mg | Rosu 20 mg + Eze 10 mg | Simva 40 mg + Eze 10 mg | Simva 80 mg + Eze 10 mg
Anaemia (Blood and lymphatic system disorders) | 0/213 | 0/212 | 0/199 | 0/203 | 0/200 | 0/191 | 0/189 | 1/192
Acute myocardial infarction (Cardiac disorders) | 0/213 | 1/212 | 0/199 | 0/203 | 0/200 | 0/191 | 0/189 | 0/192
Angina pectoris (Cardiac disorders) | 1/213 | 0/212 | 0/199 | 0/203 | 1/200 | 0/191 | 0/189 | 0/192
Angina unstable (Cardiac disorders) | 0/213 | 0/212 | 0/199 | 0/203 | 2/200 | 0/191 | 3/189 | 0/192
Cardiac failure (Cardiac disorders) | 0/213 | 1/212 | 0/199 | 0/203 | 0/200 | 0/191 | 0/189 | 0/192
Myocardial ischaemia (Cardiac disorders) | 0/213 | 0/212 | 0/199 | 0/203 | 0/200 | 0/191 | 1/189 | 0/192
Ventricular extrasystoles (Cardiac disorders) | 0/213 | 1/212 | 0/199 | 0/203 | 0/200 | 0/191 | 0/189 | 0/192
Liver disorder (Hepatobiliary disorders) | 0/213 | 0/212 | 0/199 | 1/203 | 0/200 | 0/191 | 0/189 | 0/192
Abdominal abscess (Infections and infestations) | 0/213 | 0/212 | 0/199 | 0/203 | 0/200 | 0/191 | 0/189 | 1/192
Diverticulitis (Infections and infestations) | 0/213 | 0/212 | 0/199 | 0/203 | 0/200 | 0/191 | 0/189 | 1/192
Pneumonia (Infections and infestations) | 1/213 | 0/212 | 0/199 | 0/203 | 0/200 | 0/191 | 0/189 | 0/192
Staphylococcal abscess (Infections and infestations) | 0/213 | 0/212 | 0/199 | 0/203 | 0/200 | 1/191 | 0/189 | 0/192
Fracture displacement (Injury, poisoning and procedural complications) | 0/213 | 0/212 | 0/199 | 0/203 | 0/200 | 0/191 | 1/189 | 0/192
Hypoglycaemia (Metabolism and nutrition disorders) | 0/213 | 0/212 | 0/199 | 0/203 | 0/200 | 0/191 | 0/189 | 1/192
Myopathy (Musculoskeletal and connective tissue disorders) | 0/213 | 0/212 | 0/199 | 1/203 | 0/200 | 0/191 | 0/189 | 0/192
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/213 | 0/212 | 0/199 | 0/203 | 1/200 | 0/191 | 0/189 | 0/192
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/213 | 0/212 | 0/199 | 0/203 | 0/200 | 0/191 | 1/189 | 0/192
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/213 | 0/212 | 0/199 | 0/203 | 0/200 | 0/191 | 1/189 | 0/192
Cerebral ischaemia (Nervous system disorders) | 0/213 | 0/212 | 0/199 | 1/203 | 0/200 | 0/191 | 0/189 | 0/192
Cerebrovascular accident (Nervous system disorders) | 0/213 | 2/212 | 0/199 | 0/203 | 0/200 | 0/191 | 0/189 | 0/192
Transient ischaemic attack (Nervous system disorders) | 0/213 | 0/212 | 1/199 | 0/203 | 1/200 | 0/191 | 0/189 | 0/192
Alcoholism (Psychiatric disorders) | 0/213 | 0/212 | 0/199 | 1/203 | 0/200 | 0/191 | 0/189 | 0/192
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/213 | 0/212 | 0/199 | 0/203 | 0/200 | 0/191 | 0/189 | 0/192
Arterial thrombosis limb (Vascular disorders) | 1/213 | 0/212 | 0/199 | 0/203 | 0/200 | 0/191 | 0/189 | 0/192
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Simvastatin 40 mg | Simvastatin 80 mg | Rosu 10 mg + Eze 10 mg | Rosu 20 mg + Eze 10 mg | Simva 40 mg + Eze 10 mg | Simva 80 mg + Eze 10 mg
Nausea (Gastrointestinal disorders) | 4/213 | 5/212 | 1/199 | 1/203 | 1/200 | 3/191 | 2/189 | 1/192
Oedema peripheral (General disorders) | 0/213 | 0/212 | 0/199 | 0/203 | 1/200 | 0/191 | 2/189 | 4/192
Bronchitis (Infections and infestations) | 1/213 | 1/212 | 4/199 | 2/203 | 3/200 | 2/191 | 2/189 | 1/192
Influenza (Infections and infestations) | 2/213 | 1/212 | 4/199 | 1/203 | 0/200 | 4/191 | 3/189 | 0/192
Nasopharyngitis (Infections and infestations) | 3/213 | 3/212 | 4/199 | 3/203 | 2/200 | 5/191 | 2/189 | 3/192
Upper respiratory tract infection (Infections and infestations) | 1/213 | 1/212 | 4/199 | 3/203 | 2/200 | 1/191 | 3/189 | 2/192
Arthralgia (Musculoskeletal and connective tissue disorders) | 5/213 | 4/212 | 1/199 | 4/203 | 2/200 | 0/191 | 1/189 | 2/192
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1/213 | 2/212 | 4/199 | 1/203 | 2/200 | 1/191 | 3/189 | 3/192
Myalgia (Musculoskeletal and connective tissue disorders) | 5/213 | 10/212 | 3/199 | 7/203 | 4/200 | 5/191 | 4/189 | 3/192
Dizziness (Nervous system disorders) | 1/213 | 5/212 | 1/199 | 2/203 | 1/200 | 2/191 | 3/189 | 2/192
Headache (Nervous system disorders) | 4/213 | 4/212 | 5/199 | 4/203 | 3/200 | 1/191 | 1/189 | 2/192

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No